CLINICAL TRIAL: NCT02910271
Title: Clinical Features and Prevalence of Asymptomatic Peripheral Artery Disease in Patients With Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Other Study IDs: PI464/15
Record Dates: First submitted 2016-08-10; First posted 2016-09-22 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2018-07

CONDITIONS: Type 1 Diabetes Mellitus; Peripheral Artery Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
AIMS: Determining the clinical features and prevalence of peripheral artery disease (PAD) in asymptomatics patients with type 1 diabetes mellitus (T1DM) and checking the validity of the current recommendations regarding for PAD screening in T1DM.

METHODOLOGY: An observational and cross-sectional prevalence study. The whole group of patients (sample size calculated: 299 patients) will make the Edinburgh Questionnaire for detecting classic symptoms of intermittent claudication, and after verifying the absence of symptoms and exclusion criteria, they will be included in the study. All patients will undergo assessment of clinical parameters related to T1DM and classic cardiovascular risk factors, as well as, an analytical assessment of the lipid profile, HbA1c level, proinflammatory profile and oxidative stress status. They will also undergo a comprehensive anthropometric assessment including office blood pressure (BP) monitoring and ambulatory 24-hours BP monitoring in patients with an indication as routine clinical practice, assessment of cardioautonomic function, and lastly an ankle-brachial index (ABI) by Doppler ultrasound, in the context of routine clinical practice in patients with clinical indication, or as an extraordinary procedure for participating in the study in patients who do not meet criteria for screening according to current recommendations.

DETAILED DESCRIPTION:
INTRODUCTION:

PAD is a condition characterized by atherosclerotic occlusive disease of the lower extremities. While PAD is a major risk factor for lower-extremity amputation, it is also accompanied by a high likelihood for symptomatic cardiovascular and cerebrovascular disease.

PAD is often more subtle in its presentation in patients with diabetes than in those without diabetes. In contrast to the focal and proximal atherosclerotic lesions of PAD found typically in other high-risk patients, in diabetic patients the lesions are more likely to be more diffuse and distal. Importantly, PAD in individuals with diabetes is usually accompanied by peripheral neuropathy with impaired sensory feedback, thus a classic history of claudication may be less common. Data from Framingham Heart Study revealed that 20% of PAD symptomatic patients had diabetes mellitus, but probably, this data greatly underestimates PAD prevalence. As well, it has been reported that of those with PAD, over one-half of patients are asymptomatic or have atypical symptoms, about one-third have claudication, and the rest have more severe disease. Also, patients with diabetes who have been identified with PAD are more prone to sudden ischemia secondary to arterial thrombosis or to have a pivotal event leading to neuroischemic ulceration or infection that rapidly results in an acute presentation with critical limb ischemia and risk of amputation.

However, is important to note, that most clinical data about PAD and diabetes, are becoming from population studies and randomized clinical trials, made up exclusively with type 2 patients, or more frequently, after analyzing all patients with diabetes diagnosis, without distinction between T1 to T2 subtypes. Thus, although much is known regarding PAD in the general population, the assessment and management of PAD in those with diabetes is less clear, especially in patients with T1DM diagnosis.

In 2003, a Consensus Development Conference was held regarding PAD in diabetes. After a series of lectures by experts in the field of endocrinology, cardiology, vascular surgery, orthopedic surgery, podiatry, and nursing, a vascular medicine panel was asked to answer questions about the epidemiology and impact of PAD in people with diabetes, diagnosis and treatment of PAD, but always generalizing the management of T1 and T2 diabetes, under the unique same term of "diabetes".

PAD diagnosing in patients with diabetes is of clinical importance for two reasons:

i) to identify patients at high risk of subsequent cardiovascular and cerebrovascular disease ii) to diagnose and treat PAD, which may be associated with functional disability and limb loss.

Preventive measures in a patient with subclinical disease will make possible to avoid acute and chronic complications. Therefore, the knowledge about the true prevalence of PAD in T1DM is relevant for setting the screening indication in this patients, given that this is frequently asymptomatic and it might be clinically different at presentation compared to type 2 diabetes patients.

AIMS:

The main objective of this works is determine the clinical features and prevalence of PAD in asymptomatics patients with T1DM and check the validity of the current recommendations regarding for PAD screening in T1DM.

METHODOLOGY:

Observational and cross-sectional prevalence study will be conducted. A consecutive population of type 1 patients from our clinics (sample size calculated: 299 patients) will be screened by the Edinburgh Questionnaire (Leng & Fowkes 1992) for detecting classic symptoms of intermittent claudication, and after verifying the absence of symptoms and exclusion criteria, they will be included in the study.

* All patients will undergo assessment of clinical parameters related to T1DM (years of the initial diagnosis, insulin treatment, metabolic control, microvascular chronic complications), cardiovascular risk factors (hypertension, dyslipidemia, chronic smoking), prior cardiovascular disease (coronary and cerebrovascular disease), as well as, an analytical assessment including a lipid profile, HbA1c level, proinflammatory markers (C-reactive protein, homocysteine) and oxidative stress status.
* They will undergo a comprehensive anthropometric evaluation: weight, height, body mass index [BMI (kg / m2)], abdominal and hip circumference, and body fat percentage to total body weight by bioelectrical impedance.
* Office BP and ambulatory 24-hours BP monitoring in patients with an indication as routine clinical practice (Mancia G. et al 2013).
* Assessment of cardiovascular autonomic dysfunction: orthostatism systolic and diastolic BP, orthostatism heart rate, heart rate variability to expiration / inspiration, Valsalva and orthostatic.
* Diabetic foot exploration (including bilateral peripheral pulses, Neuropathy Symptoms Score questionnaire, monofilament exploration, and calibrated tuning fork).
* The ABI will be performed by Doppler ultrasound (HADECO® Minidop 8 Mhz), in the context of routine clinical practice in patients with clinical indication, or an extraordinary procedure for participating in the study in patients who do not meet criteria for screening according to current recommendations.

The ABI will be measured in both posterior tibial and pedia arteries. Interpretation of ABI wil be as follows: Average: 0.90 to 1.20; mild arterial obstruction: 0.70 to 0.89; moderate arterial obstruction: 0.40 to 0.69; severe arterial obstruction < 0.40; poorly compressible arteries > 1.20.

In patients with ABI > 1.20 or < 0.9, the examination will be completed as recommended guidelines about asymptomatic PAD diagnosis by assessing the graphic recording blood flow and assessment index finger-arm.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of T1DM before 30 years of age.

DM diagnostic criteria:

* DM cardinal symptoms (polyuria, polydipsia, unexplained weight loss) with plasma glucose ≥ 200 mg / dl, or diagnosis as diabetic ketoacidosis (DKA).
* fasting plasma glucose (≥ 8 h) ≥ 126 mg / dl.
* plasma glucose at 2 h in testing oral glucose tolerance test (75 g glucose) ≥ 200 mg / dl.
* glycosylated hemoglobin (HbA1c) ≥ 6.5% [as certified by the National method Glycohemoglobin Standardized Program (NGSP) and standardized according to the Diabetes Control and Complication Trial trial (DCCT)].

The criteria b, c and d require confirmation, except in cases of hyperglycemia with acute decompensation (criteria a).

* Positive determination of a autoantibody serum markers of immune destruction against antigens cytoplasm of the islet cells (ICA), anti-insulin (AAI), and / or anti protein glutamate decarboxylase (GADA) at initial diagnosis time or during the course of the disease.

Acceptance of participation in the study and sign the informed consent.

Exclusion Criteria:

* Prior diagnosis of PAD, diabetic foot, leg amputation or symptoms in line with PAD according to the Edinburgh questionnaire for intermittent claudication.
* Diagnosis of type 2 diabetes, gestational diabetes, latent autoimmune diabetes in adults (LADA) or maturity-onset diabetes of youth (MODY) diabetes.
* Current pregnancy, institutionalized or terminal illness subjects.
* Refusal to participate in the study or to sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prior diagnosis of T1DM ≥ 18 years old, consecutively selected from T1DM and Insulin Pump clinics of a tertiary Hospital in Madrid.
Sampling Method: Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of PAD in asymptomatic patients with T1DM assessed by ankle-branchial index. | 2 years

SECONDARY OUTCOMES:
Association between anthropometric parameters and asymptomatic peripheral artery disease in patients with type 1 diabetes mellitus. | 2 years
  Comparison of anthropometric parameters among patients with and without peripheral artery disease.
  Anthropometric evaluation includes:
  * Body mass index.
  * Waist circumference.
  * Body fat percentage with respect to total body weight assessed by bioelectrical impedance.
Association between lipid profile and asymptomatic artery disease in patients with type 1 diabetes mellitus. | 2 years
  Comparison of lipids among patients with and without peripheral artery disease.
  Lipid profile includes:
  * Total cholesterol.
  * LDL-cholesterol.
  * HDL-cholesterol.
  * Triglycerides.
  * Total cholesterol / HDL-cholesterol.
  * NonHDL cholesterol.
Association between glycemic control and asymptomatic artery disease in patients with type 1 diabetes mellitus. | 2 years
  Comparison of glycosylated hemoglobin levels among patients with and without peripheral artery disease.
Association between C-reactive protein and asymptomatic artery disease in patients with type 1 diabetes mellitus. | 2 years
  Comparison of circulating C-reactive protein among patients with and without peripheral artery disease.
Association between homocysteine and asymptomatic artery disease in patients with type 1 diabetes mellitus. | 2 years
  Comparison of circulating homocysteine levels among patients with and without peripheral artery disease.
Number and percentage of patients with pathological ankle-branchial index without screening criteria according to the current recommendations for subjects with type 1 diabetes mellitus. | 2 years
  Comparison of ankle-branchial index by doppler technique among patients with and without screening criteria according to the current recommendations for subjects with type 1 diabetes mellitus.
Number and percentage of patients with type 1 diabetes mellitus, cardiovascular autonomic dysfunction and asymptomatic PAD. | 2 years
  Cardiovascular autonomic dysfunction will be assessed by orthostatism induced abnormal changes in systolic BP and diastolic BP.
Number and percentage of patients with type 1 diabetes mellitus, cardiovascular autonomic dysfunction and asymptomatic PAD. | 2 years
  Cardiovascular autonomic dysfunction will be assessed by orthostatism induced abnormal changes in heart rate.
Number and percentage of patients with type 1 diabetes mellitus, cardiovascular autonomic dysfunction and asymptomatic PAD. | 2 years
  Cardiovascular autonomic dysfunction will be assessed by RR interval variability response to expiration / inspiration, Valsalva maneuver and orthostatism.
Prevalence of asymptomatic atherosclerotic carotid disease in patients with asymptomatic PAD. | 2 years
  Asymptomatic carotid atherosclerotic disease will be assessed by measuring the thickness of the intima by doppler technique.

CONTACTS AND LOCATIONS:
Overall Officials: María Lía Nattero Chávez, Principal Investigator — Diabetes, Obesity and Human Reproduction Research Group, Department of Endocrinology and Nutrition, Hospital Universitario Ramón y Cajal, Universidad de Alcalá, Instituto Ramón y Cajal de Investigación Sanitaria (IRYCIS)
Locations (1):
- Diabetes, Obesity and Human Reproduction Research Group, Department of Endocrinology and Nutrition, Hospital Universitario Ramón y Cajal, Universidad de Alcalá, Instituto Ramón y Cajal de Investigación Sanitaria (IRYCIS), Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Ferranti SD, de Boer IH, Fonseca V, Fox CS, Golden SH, Lavie CJ, Magge SN, Marx N, McGuire DK, Orchard TJ, Zinman B, Eckel RH. Type 1 diabetes mellitus and cardiovascular disease: a scientific statement from the American Heart Association and American Diabetes Association. Circulation. 2014 Sep 23;130(13):1110-30. doi: 10.1161/CIR.0000000000000034. Epub 2014 Aug 11. No abstract available. PMID 25114208
- [Background] American Diabetes Association. Peripheral arterial disease in people with diabetes. Diabetes Care. 2003 Dec;26(12):3333-41. doi: 10.2337/diacare.26.12.3333. No abstract available. PMID 14633825
- [Background] Murabito JM, D'Agostino RB, Silbershatz H, Wilson WF. Intermittent claudication. A risk profile from The Framingham Heart Study. Circulation. 1997 Jul 1;96(1):44-9. doi: 10.1161/01.cir.96.1.44. PMID 9236415
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Halperin JL, Hiratzka LF, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery; Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines; American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; Vascular Disease Foundation. ACC/AHA 2005 guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): executive summary a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease) endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. J Am Coll Cardiol. 2006 Mar 21;47(6):1239-312. doi: 10.1016/j.jacc.2005.10.009. No abstract available. PMID 16545667
- [Background] Standards of Medical Care in Diabetes-2016: Summary of Revisions. Diabetes Care. 2016 Jan;39 Suppl 1:S4-5. doi: 10.2337/dc16-S003. No abstract available. PMID 26696680
- [Background] Leng GC, Fowkes FG. The Edinburgh Claudication Questionnaire: an improved version of the WHO/Rose Questionnaire for use in epidemiological surveys. J Clin Epidemiol. 1992 Oct;45(10):1101-9. doi: 10.1016/0895-4356(92)90150-l. PMID 1474406
- [Background] Parati G, Stergiou G, O'Brien E, Asmar R, Beilin L, Bilo G, Clement D, de la Sierra A, de Leeuw P, Dolan E, Fagard R, Graves J, Head GA, Imai Y, Kario K, Lurbe E, Mallion JM, Mancia G, Mengden T, Myers M, Ogedegbe G, Ohkubo T, Omboni S, Palatini P, Redon J, Ruilope LM, Shennan A, Staessen JA, vanMontfrans G, Verdecchia P, Waeber B, Wang J, Zanchetti A, Zhang Y; European Society of Hypertension Working Group on Blood Pressure Monitoring and Cardiovascular Variability. European Society of Hypertension practice guidelines for ambulatory blood pressure monitoring. J Hypertens. 2014 Jul;32(7):1359-66. doi: 10.1097/HJH.0000000000000221. PMID 24886823
- [Background] Nattero-Chavez L, Redondo Lopez S, Alonso Diaz S, Garnica Urena M, Fernandez-Duran E, Escobar-Morreale HF, Luque-Ramirez M. Association of Cardiovascular Autonomic Dysfunction With Peripheral Arterial Stiffness in Patients With Type 1 Diabetes. J Clin Endocrinol Metab. 2019 Jul 1;104(7):2675-2684. doi: 10.1210/jc.2018-02729. PMID 30786000
- [Background] Nattero-Chavez L, Alonso Diaz S, Jimenez-Mendiguchia L, Garcia-Cano A, Fernandez-Duran E, Dorado Avendano B, Escobar-Morreale HF, Luque-Ramirez M. Sexual Dimorphism and Sex Steroids Influence Cardiovascular Autonomic Neuropathy in Patients With Type 1 Diabetes. Diabetes Care. 2019 Nov;42(11):e175-e178. doi: 10.2337/dc19-1375. Epub 2019 Sep 17. No abstract available. PMID 31530659
- [Background] Nattero-Chavez L, Bayona Cebada A, Fernandez-Duran E, Quintero Tobar A, Dorado Avendano B, Escobar-Morreale H, Luque-Ramirez M. "Arterial stiffness is not associated with changes in the circadian pattern of blood pressure in patients with type 1 diabetes mellitus and cardiovascular autonomic dysfunction". Diab Vasc Dis Res. 2023 May-Jun;20(3):14791641231173621. doi: 10.1177/14791641231173621. PMID 37184151
- [Result] Nattero-Chavez L, Luque-Ramirez M, Moncayo S, Alonso-Diaz S, Fernandez-Duran E, Redondo-Lopez S, Garcia-Urena M, Escobar-Morreale HF. Circulating soluble klotho is not associated with an elevated ankle-brachial index as a surrogate marker of early arterial calcification in patients with type 1 diabetes mellitus and no evidence of renal dysfunction. Diabetes Metab. 2019 Dec;45(6):589-592. doi: 10.1016/j.diabet.2018.01.009. Epub 2018 Jan 18. No abstract available. PMID 29398255
- [Result] Nattero-Chavez L, Redondo Lopez S, Alonso Diaz S, Garnica Urena M, Fernandez-Duran E, Escobar-Morreale HF, Luque-Ramirez M. The peripheral atherosclerotic profile in patients with type 1 diabetes warrants a thorough vascular assessment of asymptomatic patients. Diabetes Metab Res Rev. 2019 Feb;35(2):e3088. doi: 10.1002/dmrr.3088. Epub 2018 Nov 20. PMID 30338903
- [Result] Nattero-Chávez L, Alonso Díaz S, Montanez L, Fernández E, Redondo López S, Garnica Ureña M, Bayona A, Esxobar-Morreale HF, Luque-Ramírez M. 567-P: Influence of Sex on Cardioautonomic Neuropathy in Patients with Type 1 Diabetes. Diabetes 2019 Jun; 68(Supplement 1): -. https://doi.org/10.2337/db19-567-P
- [Result] Nattero-Chavez L, Martinez-Garcia MA, Fernandez-Duran E, Redondo Lopez S, Dorado Avendano B, Escobar-Morreale HF, Luque-Ramirez M. Fasting serum copeptin and asymptomatic peripheral artery disease: No association in patients with type 1 diabetes mellitus. Diabetes Metab. 2021 May;47(3):101207. doi: 10.1016/j.diabet.2020.10.005. Epub 2020 Nov 4. PMID 33160031
- [Result] Nattero-Chavez L, Martinez-Garcia MA, Redondo Lopez S, Fernandez-Duran E, Dorado Avendano B, Escobar-Morreale HF, Luque-Ramirez M. High serum copeptin may be a marker of an increased carotid intima-media thickness in asymptomatic patients with type 1 diabetes. J Diabetes Complications. 2022 Jan;36(1):108085. doi: 10.1016/j.jdiacomp.2021.108085. Epub 2021 Nov 11. PMID 34823978